CLINICAL TRIAL: NCT01482819
Title: Evaluation of Daytime Corneal Swelling During Wear of Galyfilcon A Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CR-005031
Record Dates: First submitted 2011-11-16; First posted 2011-12-01 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (10):
- Sequence 1 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Lotrafilcon A
  2. Spectacles
  3. Galyfilcon A Plus
  4. Polymacon
  5. Galyfilcon A
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 2 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Galyfilcon A Plus
  2. Galyfilcon A
  3. Lotrafilcon A
  4. Polymacon
  5. Spectacles
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 3 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Galyfilcon A
  2. Polymacon
  3. Galyfilcon A Plus
  4. Spectacles
  5. Lotrafilcon A
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 4 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Spectacles
  2. Lotrafilcon A
  3. Polymacon
  4. Galyfilcon A Plus
  5. Galyfilcon A
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 5 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Polymacon
  2. Galyfilcon A
  3. Spectacles
  4. Galyfilcon A Plus
  5. Lotrafilcon A
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 6 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Galyfilcon A
  2. Galyfilcon A Plus
  3. Polymacon
  4. Lotrafilcon A
  5. Spectacles
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 7 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Polymacon
  2. Spectacles
  3. Galyfilcon A
  4. Lotrafilcon A
  5. Galyfilcon A Plus
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 8 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Galyfilcon A Plus
  2. Lotrafilcon A
  3. Galyfilcon A
  4. Spectacles
  5. Polymacon
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 9 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Lotrafilcon A
  2. Galyfilcon A Plus
  3. Spectacles
  4. Galyfilcon A
  5. Polymacon
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles
- Sequence 10 (Other): Five separate sessions of bilateral lens wear of 8 to 12 hours; each session separated by a minimum of 24 hours. This sequence is as follows:
  1. Spectacles
  2. Polymacon
  3. Lotrafilcon A
  4. Galyfilcon A
  5. Galyfilcon A Plus
  Interventions: Device: galyfilcon A; Device: galyfilcon A plus; Device: lotrafilcon A; Device: polymacon; Other: spectacles

INTERVENTIONS:
Device: galyfilcon A — contact lenses worn bilaterally for 8-12 hours
Device: galyfilcon A plus — contact lenses worn bilaterally for 8-12 hours
Device: lotrafilcon A — contact lenses worn bilaterally for 8-12 hours
Device: polymacon — contact lenses worn bilaterally for 8-12 hours
Other: spectacles — habitual spectacles owned by subject, non-specific manufacturer

SUMMARY:
The purpose of this study is to evaluate corneal swelling, limbal redness, and endothelial bleb response to wearing galyfilcon A lenses in asian eyes.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age (i.e. 18 years)
* Be of Asian descent and have -Asian eye‖ identifying features (see Appendix A)
* Be mentally competent, willing and able to sign a written informed consent form.
* Have contact lens distance sphere requirement in the range 1.00D to 6.00D.
* Have spectacle astigmatism <1.25D in each eye
* Currently wear soft contact lenses (for at least 3 months prior to the trial ) without experiencing difficulties or contact lens related complications
* Have had an oculo-visual examination within the previous 12 months.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  * No evidence of lid abnormality or infection
  * No conjunctival abnormality or infection
  * No clinically significant slit lamp findings (i.e. edema, staining, scarring, vascularization, infiltrates or abnormal opacities)
  * No other active ocular disease

Exclusion Criteria:

* Requires concurrent ocular medication.
* Clinically significant (Grade 3 or 4) corneal staining (FDA scale), corneal stromal haze, corneal vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Has had refractive surgery.
* Has had any anterior ocular surgery. Has had any other ocular surgery or injury within 8 weeks immediately prior to enrolment for this study.
* History of abnormal lachrymal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Extended lens wear in last 3 months.
* PMMA, hybrid or RGP lens wear in the previous 8 weeks
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Has diabetes
* Known/reported infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* History of chronic eye disease (e.g. glaucoma or ARMD).
* Pregnancy, lactating, or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial or in last 30 days.
* Family member or employee of the clinical site, investigator or other study staff.
* Currently wears habitual contact lenses on an EW basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hawthorn, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Twenty-one subjects were enrolled, and 19 subjects completed the study per protocol. Two subjects were discontinued. There were no ineligible subjects.
Period: Overall Study
Arm/Group | All Subjects
Started | 21
Completed | 19
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Subjects who were screened, gave consent, enrolled, and were randomized in the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5
  Multiple | 16
Region of Enrollment [Number; unit: participants]
  Australia | 21

OUTCOME MEASURES:

1. Primary Outcome: Corneal Swelling
Description: measured in microns using the Optical Low Coherence Reflectometry (OLCR) Pachymeter. This pachymeter gives corneal thickness measurements to the accuracy of 1 micron (µm)
Time Frame: after 8 hours of lens wear
Population: Subjects who were enrolled, randomized, and completed the study. One eye from each subject was measured.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Groups:
- Spectacles: No lenses, glasses wear only, testing is done on open eye once glasses are removed. Acted as a negative control.
- Galyfilcon A Plus; Galyfilcon A; Lotrafilcon A; Polymacon: Test article
Arm/Group | Spectacles | Galyfilcon A Plus | Galyfilcon A | Lotrafilcon A | Polymacon
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19
Number analyzed (eyes) | 19 | 19 | 19 | 19 | 19
microns | 569.42 (36.0709) | 574.64 (39.7804) | 575.57 (37.6229) | 578.99 (41.4960) | 573.79 (36.1644)

2. Primary Outcome: Limbal Redness
Description: grade scale of 0 to 4, where 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe; reported as an average grade.
Time Frame: after 8 hours of lens wear
Population: Subjects who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Spectacles | Galyfilcon A Plus | Galyfilcon A | Lotrafilcon A | Polymacon
Number analyzed (Participants) | 19 | 19 | 20 | 20 | 19
Number analyzed (eyes) | 38 | 38 | 40 | 40 | 38
units on a scale | 0.66 (0.2479) | 0.83 (0.3023) | 0.77 (0.3085) | 0.91 (0.3087) | 1.14 (0.3363)

3. Primary Outcome: Endothelia Blebs
Description: 0 to 100% of area; measured as a percentage of corneal area with blebs.
Time Frame: after 20 minutes of lens wear
Population: Subjects who were enrolled, randomized and completed the study.
Measure: Mean (Standard Deviation); unit: percentage of area
Units Other Than Participants: eyes
Arm/Group | Spectacles | Galyfilcon A Plus | Galyfilcon A | Lotrafilcon A | Polymacon
Number analyzed (Participants) | 20 | 19 | 20 | 20 | 19
Number analyzed (eyes) | 40 | 38 | 40 | 40 | 38
percentage of area | 4.97 (3.3703) | 8.86 (3.9396) | 10.93 (6.6020) | 10.31 (6.6747) | 8.50 (3.6000)

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less